CLINICAL TRIAL: NCT05131893
Title: Neoadjuvant Treatment of Breast Cancer - a Prospective Observational Study, PANnon ONCology (PANONC) Group Non-commercial Clinical Trial
Brief Title: Neoadjuvant Treatment of Breast Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: National Institute of Oncology, Hungary (Other)
Responsible Party: Principal Investigator, Dr. Zoltan Matrai, Head of Surgical Oncology, National Institute of Oncology, Hungary
Other Study IDs: PANONC-1 Version: 1.1
Record Dates: First submitted 2021-07-30; First posted 2021-11-23 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Breast Cancer
Keywords: Neoadjuvant systemic therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen; Goserelin; Letrozole; Epirubicin; Cyclophosphamide; Docetaxel; Paclitaxel; Trastuzumab; pertuzumab; Capecitabine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- LuminalA: 1. tamoxifen (+ LHRH analogue for premenopausal participant)
  2. non-steroidal aromatase inhibitor (+ LHRH analogue for premenopausal participant)
  3. Non-steroidal aromatase inhibitor in non-resectable tumor (+ LHRH analogue in premenopausal participant) + CDK4 / 6 inhibitor
  Interventions: Drug: Tamoxifen; Drug: Goserelin; Drug: Letrozole 2.5Mg Tab
- LuminalB (Her2 negative): 1. 12 times weekly paclitaxel (80 mg / m˄2) followed by 4 times every 3 weeks epirubicin (E) (90-100 mg / m˄2) + cyclophosphamide (C) (600) (preferred)
  2. 4x 3 weekly E (90-100mg / m˄2) + C (600mg / m˄2), then
     1. docetaxel (90-100 mg / m˄2) 4 times in every 3 weeks or
     2. 12x weekly paclitaxel (80mg / m˄2)
  3. 4x every 2 weeks Epirubicin (E) (90-100mg / m˄2) + Cyclophosphamid (C) (600mg / m˄2), then
     1. 4 times every 2 weeks with paclitaxel (175 mg / m˄2) or
     2. 12x weekly paclitaxel (80mg / m˄2)
  4. TC: docetaxel (75 mg / m˄2) + cyclophosphamide (600 mg / m˄2) every 21 days with GCSF prevention (6 cycles)
  Interventions: Drug: Tamoxifen; Drug: Goserelin; Drug: Letrozole 2.5Mg Tab; Drug: Epirubicin; Drug: cyclophosphamide; Drug: Docetaxel; Drug: paclitaxel; Drug: trastuzumab
- Her2 positive: 1. 4x 3 weeks E (90-100mg / m˄2) + C (600mg / m˄2), then
     1. 12 times weekly paclitaxel + trastuzumab (every week or 3 weekly) +/- pertuzumab (3 weekly) or
     2. 4x 3 weekly docetaxel (100mg / m˄2) + trastuzumab +/- pertuzumab
  2. Docetaxel (75 mg / m˄2) + carboplatin (AUC6) + trastuzumab +/- pertuzumab 6 times every 3 weeks c) E (90-100mg / m˄2) + C (600mg / m˄2) 4x every 2 weeks, then 12 times weekly paclitaxel + trastuzumab (every week or 3 weekly) +/- pertuzumab (3 weekly)
  Interventions: Drug: Tamoxifen; Drug: Goserelin; Drug: Letrozole 2.5Mg Tab; Drug: Epirubicin; Drug: cyclophosphamide; Drug: Docetaxel; Drug: paclitaxel; Drug: trastuzumab; Drug: pertuzumab
- Triple-negative breast cancer: 1. Paclitaxel (80 mg / m˄2) +/- carboplatin (AUC2) 12 times weekly, then E (90-100 mg / m˄2) + C (600 mg / m˄2) 4 times three weekly (preferred)
  2. 4x every 3 weeks E (90-100mg / m˄2) + C (600mg / m˄2), then
     1. 4x docetaxel (90-100mg / m˄2) or
     2. 12x weekly paclitaxel (80mg / m˄2) +/- carboplatin (AUC2 )
  3. 4x every 2 weeks E (90-100mg / m˄2) + C (600mg / m˄2), then
     1. 4 times every 2 weeks paclitaxel (175 mg / m˄2) or
     2. 12x weekly paclitaxel (80mg / m˄2) +/- carboplatin (AUC2)
  Interventions: Drug: Epirubicin; Drug: cyclophosphamide; Drug: Docetaxel; Drug: paclitaxel; Drug: Capecitabine

INTERVENTIONS:
Drug: Tamoxifen — endocrine therapy
  Groups: Her2 positive; LuminalA; LuminalB (Her2 negative)
Drug: Goserelin — endocrine therapy
  Groups: Her2 positive; LuminalA; LuminalB (Her2 negative)
Drug: Letrozole 2.5Mg Tab — endocrine therapy
  Other Names: letrozole
  Groups: Her2 positive; LuminalA; LuminalB (Her2 negative)
Drug: Epirubicin — chemotherapy
  Groups: Her2 positive; LuminalB (Her2 negative); Triple-negative breast cancer
Drug: cyclophosphamide — chemotherapy
  Groups: Her2 positive; LuminalB (Her2 negative); Triple-negative breast cancer
Drug: Docetaxel — chemotherapy
  Groups: Her2 positive; LuminalB (Her2 negative); Triple-negative breast cancer
Drug: paclitaxel — chemotherapy
  Groups: Her2 positive; LuminalB (Her2 negative); Triple-negative breast cancer
Drug: trastuzumab — biological treatment
  Groups: Her2 positive; LuminalB (Her2 negative)
Drug: pertuzumab — biological treatment
  Groups: Her2 positive
Drug: Capecitabine — chemotherapy
  Groups: Triple-negative breast cancer

SUMMARY:
Observational investigation of participants who are given neoadjuvant treatment for invasive breast cancer. The scope of the study is to collect information on standardized treatment results, to explore the causes of dose modification and its effect on efficacy, to explore potential prognostic factors, and to explore the long-term side effects of different treatment modalities.

DETAILED DESCRIPTION:
The purpose of the study is based on the uniform application of international guidelines in Hungarian conditions. The standardized circumstances may lead to optimization of neoadjuvant therapy, it may facilitate subsequent data analysis, provide a basis for prospective clinical questions, and demonstrate improvement in pathologic complete remission (pCR) and overall survival (OS) compared to historical control. It may make possible to collect real-life data on each therapeutic option: efficacy, side effects, dose reduction, dose intensity, long-term consequences. The main scope is to collect prospective data to explore prognostic and predictive factors. The auxiliary aim is the assessment and comparison of quality of life during specific treatments and their side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Participant over 18 years of age .
2. Histologically confirmed (core biopsy) invasive breast tumor.
3. Tumor extent for the indication:

   * regression must be achieved for radical surgical removal or
   * regression is required for breast-conserving surgery or
   * if hormone receptor (HR)-positive and Her2-: stage IIB (cT2N1 or cT3NO) - IIIC,
   * if HR-negative: stage IIA (cT2N0 or cT0-1N1) - IIIC Note: In the case of a locally advanced, irresectable case, if the possibility of radical surgery later is a realistic goal, the participant may be included in the study.
4. Appropriate general condition: ECOG 0-1
5. Proper organ function

   * Neutrophil count ≥ 1.5 G / l, platelet count ≥ 100 G / l, hemoglobin ≥ 10 g / dl
   * Alanine aminotransferase (ALT) / aspartate aminotransferase (AST) is less than 1.5 times the upper limit of the normal range
   * bilirubin less than 1.5 times the upper limit of the normal range (except Gilbert's disease, where less than 3 times)
   * creatinine less than 1.5 times the upper limit of the normal range or estimated glomerular filtration rate (eGFR) higher than 60 ml / min

Exclusion Criteria:

1. Proven or suspected distant metastasis.
2. No staging studies have been performed: at least chest x-ray, abdominal ultrasound. It is preferred to perform CT from the chest, abdomen, pelvic regions and bone isotope, or PET / CT if possible in case of lymph node involvement.
3. Known significant heart disease: major arrhythmia or significant conduction defect (grade 2 or more), infarction or unstable angina within 6 months, cardiac collapse without appropriate therapy, long QT syndrome, heart failure (≥New York Heart Association/NYHA II)
4. Other severe acute or chronic conditions (organic or psychiatric illness, laboratory abnormality) that, in the opinion of the treating physician, result in an unacceptable increase in the risk of chemotherapy and are contraindicated in routine clinical practice.
5. Pregnancy or if the participant does not agree to use an appropriate non-hormonal method of contraception.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients for whom neoadjuvant therapy is proposed by multidisciplinary team
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
pathological complete remission rate | 3 year, maximum
  no invasive tumor in breast and axilla

SECONDARY OUTCOMES:
invasive disease-free survival | 10 years
  from the beginning of neoadjuvant therapy to the first appearance of invasive tumor or death
European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) | 4 years
  Global health status, functional and symptom scales survey using the EORTC QLQ-C30 questionnaire before cycle 1, before cycle 4, after the last neoadjuvant chemotherapy, and before surgery, 1 year after chemotherapy
European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Breast Cancer Module (EORTC QLQ BR45) | 4 years
  Breast cancer-specific functional scales and symptom scales survey using the EORTC QLQ BR45 questionnaire before cycle 1, before cycle 4, after the last neoadjuvant chemotherapy, and before surgery, 1 year after chemotherapy
evaluation of side effects | 10 years
  to collect information all potential complaints and adverse event during and after treatment

OTHER OUTCOMES:
dose density assessment | 3 year, maximum
  actual dose / planned dose
investigate the potential prognostic effect of neutrophil/lymphocyte ratio | 10 years
  study of the role of neutrophil/lymphocyte ratio (NLR) at baseline, before the 3. cycle, and before surgery. NLR is measured from the qualitative blood count as the absolute neutrophil count divided by the absolute lymphocyte count
investigate the potential prognostic effect of monocyte/lymphocyte ratio | 10 years
  monocyte/lymphocyte ratio (MLR) at baseline, before the 3. cycle, and before surgery. MLR is measured from the qualitative blood count as the absolute monocyte count divided by the absolute lymphocyte count
investigate potential prognostic factors, CRP | 10 years
  C-reactive protein serum level befor start of chemotherapy
investigate potential prognostic factors | 10 years
  circulating free-DNA at baseline, before 3. cycle, before surgery

CONTACTS AND LOCATIONS:
Overall Officials: Gabor Rubovszky, Principal Investigator — NIO Hungary
Locations (1):
- National Institute of Oncolgy, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No
The individual participant data are not planned to be shared with other researchers but will be available upon request except personal data